CLINICAL TRIAL: NCT05327673
Title: Impact of the Use of Allogeneic Hematopoietic Stem Cell Transplantation in Reunion Island Patients: Quality of Life, Determinants of Choices and Financial Repercussions
Acronym: AlloRé
Status: Not yet recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de la Réunion (Other)
Collaborators: Institut Paoli-Calmettes (Other)
Responsible Party: Sponsor
Other Study IDs: 2020/CHU/21
Record Dates: First submitted 2022-04-07; First posted 2022-04-14 (Actual); Last update posted 2022-04-21 (Actual); Status verified 2022-04

CONDITIONS: Allogeneic Hematopoietic Stem Cell Transplantation
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients who accept Allogeneic Hematopoietic Stem Cell Transplantation (alloH SCT)
  Interventions: Other: questionnaire
- patients who did not accept Allogeneic Hematopoietic Stem Cell Transplantation (alloH SCT)
  Interventions: Other: questionnaire

INTERVENTIONS:
Other: questionnaire — * quality of life score: FACT-BMT
  * decisional conflict scale
  * Discreet Choice Experiment questionnaire

SUMMARY:
This project aims to document and analyse - with a three-fold anthropological, psychosocial and economical approach - the consequences of the geographical distance from mainland France on the alloSCT on both patients, their caregivers and the healthcare system. It is organised in 3 working packages (WP).

ELIGIBILITY:
Inclusion Criteria:

* patients diagnosed with hematological malignancy (myeloid acute leukemia, lymphoid acute leukemia, non-hodgkin lymphoma, Hodgkin disease, or myelodysplasic syndrome
* candidate to an allogeneic hematopoietic stem cell transplantation in mainland France ;
* Residing in Reunion Island
* Age >18 year old;
* who accept or not allogeneic hematopoietic
* Able to complete a questionnaire

Exclusion Criteria:

* Opposition to participation and collection of their data
* Person deprived of liberty by judicial or administrative decision, and person subject to legal protection (guardianship or curators)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with myeloid acute leukemia, lymphoid acute leukemia, non-hodgkin lymphoma, Hodgkin disease, or myelodysplasic syndrome candidate to an allogeneic hematopoietic stem cell transplantation in mainland
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-07 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Quality of life Functional Assessment of Cancer Therapy - Bone Marrow Transplantation questionnaire. (FACT-BMT questionnaire) | 24 months

SECONDARY OUTCOMES:
satisfaction with decision questionnaire | 24 months
decision regret scale | 24 months
fear of recurrence questionnaire | 24 months
preferences of patients questionnaire | 24 months
cost of treatment | 24 months
  impact on patients and caregivers; impact on society

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de la Réunion, Saint-Pierre, France

IPD SHARING:
Plan to Share IPD: No